CLINICAL TRIAL: NCT02032654
Title: Duration of Antibiotic Therapy for Cellulitis (DANCE): a Randomized Controlled Trial Comparing 6 to 12 Days of Antibiotic Therapy for Patients Hospitalized With Cellulitis
Brief Title: Duration of ANtibiotic Therapy for CEllulitis
Acronym: DANCE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Budget exceeded
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, W.J. Wiersinga, MD, PhD, internist, infectious diseases specialist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL44512.018.13; 4360 (Registry Identifier: Netherlands Trial Register); 2013-002106-31 (EudraCT Number); 836011024 (Other Grant/Funding Number: Netherlands Organisation for Health Research and Development (ZonMw))
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Cellulitis; Erysipelas
Keywords: antibiotics; flucloxacillin; therapy duration; cellulitis; erysipelas; skin infections; hospital
MeSH Terms: conditions — Cellulitis; Erysipelas | interventions — Floxacillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard course (Active Comparator): Flucloxacillin (1000mg iv OR, later, 500mg capsules), every 6 hours, for 6 days, followed by: Flucloxacillin 500mg capsules, every 6 hours, for 6 days
  Interventions: Drug: Flucloxacillin
- Short course (Experimental): Flucloxacillin (1000mg iv OR, later, 500mg capsules), every 6 hours, for 6 days, followed by: Placebo (for flucloxacillin 500mg) 500mg capsules, every 6 hours, for 6 days
  Interventions: Drug: Flucloxacillin; Drug: Placebo (for flucloxacillin)

INTERVENTIONS:
Drug: Flucloxacillin
  Other Names: Floxapen
Drug: Placebo (for flucloxacillin) — Sugar capsule manufactured to mimic flucloxacillin 500mg capsules
  Arms: Short course

SUMMARY:
Cellulitis is among the most common infections leading to hospitalization, yet the optimal duration of therapy remains ill defined. Pragmatically, Dutch guidelines advise 10-14 days of antibiotics, which is the current standard of care. Recently it has been shown that antibiotic treatment for pneumonia and urinary tract infections can safely and significantly be shortened. Importantly, in an outpatient setting, treatment of uncomplicated cellulitis with 5 days of antibiotics was as effective as 10 days. We hypothesize that there is no difference in outcomes when patients hospitalized with cellulitis are treated with either a short-course (6 days) or standard-course (12 days) of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to receive intravenous antibiotics for cellulitis/erysipelas
* 18 years of age or older
* Capable of giving written informed consent, able to comply with study requirements and restrictions

Exclusion Criteria:

* Allergy for flucloxacillin, other beta-lactam antibiotics or one of the additives, or flucloxacillin induced hepatitis or liver enzyme disorders.
* Concurrent use of antibiotics for other indications
* Alternative diagnosis accounting for the clinical presentation.
* All cases involving any of the following complicating factors:

  * Use of antibiotics with Gram-positive activity for more than 4 days in the past 7 days
  * Intensive care unit admission during the last 7 days
  * Severe peripheral arterial disease (Fontaine IV)
  * Severe cellulitis necessitating surgical debridement or fascial biopsy
  * Necrotizing fasciitis
  * Periorbital or perirectal involvement
  * Surgery
  * Life expectancy less than one month
  * Risk factors associated with Gram-negative pathogens as a causative agent:

    * Chronic or macerated infra-malleolar ulcers, or infra-malleolar ulcers with previous antibiotic treatment, in patients with diabetes mellitus.
    * Neutropenia
    * Cirrhosis (Child-Pugh class B or C)
    * Intravenous drug use
    * Human or animal bite
    * Skin laceration acquired in fresh or salt open water
    * Fish fin or bone injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Part 1/2: Resolution... | day 14
  Resolution of cellulitis at day 14, defined as disappearance of warmth and tenderness at the site of infection, with substantial improvement in erythema and edema
Part 2/2: ...without relapse | day 28
  No recurrence by day 28, defined as the need for additional antibiotic therapy for cellulitis

SECONDARY OUTCOMES:
Resolution without relapse | day 28
  Other operators used to define resolution at day 14 (no fever; reduction in combined erythema/edema/warmth/tenderness score of at least 2 points, or reach 0) and relapse at day 28 (no fever; stable or further improved combined score; no new antibiotics for cellulitis)
Recurrence at day 90 | 90 days
  Recurrence of cellulitis by day 90, defined as the need for additional antibiotic therapy for cellulitis
Objective speed of recovery | Up to 90 days
  Improvement in cellulitis severity score (a 7 item scoring system, each with a score between 0-3; items are erythema, warmth, tenderness, edema, ulceration, drainage and fluctuance). Determined at day 1, day 2-3, day 5-6, day 14, and day 28
Health related Quality of Life | Up to 90 days
  Using questionnaires Dutch SF-36 and EQ-5D at day 1, day 28, and day 90
Health care resource utilisation | Up to 90 days
  Determined by total antibiotic use and effect on direct and indirect health-care associated costs, using modified versions of iMTA's Productivity Cost Questionnaire (iPCQ) and Medical Consumption Questionnaire (iMCQ). Measured at day 5-6, day 28 and day 90.
Subjective speed of recovery | Up to 90 days
  Visual Analog Scales (0-10) on pain and on swelling. Determined at day 1, day 2-3, day 5-6, day 14, day 28, and day 90
Additional antibiotic usage | Up to 90 days
  Total usage of additional antibiotics for cellulitis between the end of treatment and day 90.
Time to relapse | Up to 90 days
  Time between end of treatment and the need for additional antibiotics for cellulitis

OTHER OUTCOMES:
Cellulitis severity score subgroup analysis | up to day 28
  Analysis to see if the height of the cellulitis severity score influences outcome, using a regression analysis with interaction term for severity score.
Diabetes mellitus subgroup analysis | up to day 28
  Analysis to see if having diabetes mellitus influences outcome, using a regression analysis with interaction term for diabetes.
Per protocol analysis | up to 28 days
  Like main outcome, but the following will be included: (i) patients with treatment failure, who have received at least 24 hours of study medication, and (ii) patients with treatment success, who have received at least 80% of study medication. Treatment failure is defined as the persistence or progression of signs and symptoms of the acute process after randomization, or the inability to complete the study owing to adverse events. The response is deemed indeterminate when the patients (i) received less than 80% of the study drug for reasons other than treatment failure, (ii) acquired a concomitant infection outside of the skin requiring antibiotic treatment, (iii) were lost to follow-up, or (iv) died unrelated to the primary diagnosis.
Per protocol analysis of the "resolution without relapse" secondary outcome | up to 28 days
  Like secondary outcome, but the following will be included: (i) patients with treatment failure, who have received at least 24 hours of study medication, and (ii) patients with treatment success, who have received at least 80% of study medication. Cured is defined as above (under secondary outcome). Indeterminate is (i) receiving <80% of study drug for reasons other than unblinding/requiring new AB for cellulitis/being unable to continue due to adverse effects, (ii) acquired a concomitant infection outside of the skin requiring antibiotic treatment, (iii) were lost to follow-up, or (iv) died unrelated to the primary diagnosis. Patients who are not cured nor indeterminate are failures.
Sensitivity analyses of the "resolution without relapse" secondary outcome | up to 28 days
  Similar, but requiring further improvement of symptoms by either 1 or 2 points by day 28, instead of just stability of symptoms.
Adjustments for baseline covariates | up to day 28
  Sensitivity analysis, adjusting the primary outcome for baseline covariates

CONTACTS AND LOCATIONS:
Overall Officials: W. Joost Wiersinga, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jan M. Prins, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (11):
- Netherlands (11):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Sint Lucas Andreas Ziekenhuis, Amsterdam, North Holland
  - Slotervaartziekenhuis, Amsterdam, North Holland
  - VU university medical center, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Academic Medical Center - University of Amsterdam, Amsterdam, North Holland
  - Spaarne Gasthuis Locatie Haarlem Zuid, Haarlem, North Holland
  - Tergooi, Hilversum, North Holland
  - St. Antonius Ziekenhuis locatie Utrecht, Utrecht
  - Diakonessenhuis, Utrecht
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Cranendonk DR, Hugenholtz F, Prins JM, Savelkoul PHM, Budding AE, Wiersinga WJ; DANCE Consortium. The Skin Microbiota in Patients Hospitalized for Cellulitis and Association With Outcome. Clin Infect Dis. 2019 Apr 8;68(8):1292-1299. doi: 10.1093/cid/ciy709. PMID 30321312
- [Derived] Cranendonk DR, Opmeer BC, Prins JM, Wiersinga WJ. Comparing short to standard duration of antibiotic therapy for patients hospitalized with cellulitis (DANCE): study protocol for a randomized controlled trial. BMC Infect Dis. 2014 May 5;14:235. doi: 10.1186/1471-2334-14-235. PMID 24885384
- See also: Published study protocol in BMC Infectious Diseases — http://www.biomedcentral.com/1471-2334/14/235

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT02032654/Prot_SAP_000.pdf